CLINICAL TRIAL: NCT04244916
Title: Prospective Study to Investigate the Relevance of Monitoring Area Under the Curve of Mycophenolic Acid in Patients Receiving Mycophenolate Mofetil to Treat a Diffuse Cutaneous or a Pulmonary Involvement of Systemic Sclerosis
Brief Title: MPA AUC Monitoring in Patients Receiving MMF for Diffuse Cutaneous or Pulmonary Involvement in Systemic Sclerosis
Acronym: SCLERAMAC
Status: Terminated | Type: Observational
Why Stopped: Departure of the coordinator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190933
Record Dates: First submitted 2020-01-06; First posted 2020-01-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; diffuse; interstitial lung disease; therapeutic drug monitoring (TDM); mycophenolate mofetil
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: AUC of MPA measure — Plasmatic AUC determination of MPA requires 3 blood punctures at H0, H30 and H2.
  These punctures will be made at inclusion after 6 weeks, 12 weeks, 6 months and one year.

SUMMARY:
To define a target value of AUC MPA to improve the modified Rodnan score and / or respiratory impairment (DLCO or FVC) at one year in patients receiving MMF for the treatment of diffuse cutaneous or interstitial lung damage of systemic sclerosis.

DETAILED DESCRIPTION:
In the treatment of autoimmune diseases, MMF is almost always prescribed at a fixed dose, regardless of AUC, or based on the target of AUC determined for organ transplantation. One study looked at determining an "effective" AUC threshold in systemic lupus erythematosus, which appears to be 35mg / h / l. This was also done for ANCA vasculitis.

We therefore conducted this study to determine a correlation between AUC MPA and the effectiveness of MMF in systemic sclerosis.

Prospective, observational, open study.

Main objective: define a target value of AUC MPA to improve the modified Rodnan score and / or respiratory impairment (DLCO or FVC) at one year in patients receiving MMF for the treatment of diffuse skin involvement or pulmonary function in systemic sclerosis.

The main endpoint will be evaluated on the evolution of the modified Rodnan score at 1 year after the initiation of MMF and / or the evolution of FVC and DLCO at 1 year after the initiation of MMF.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis meeting the ACR / EULAR criteria of 2013
* Equal or more than 18 years old, able to freely consent to study
* In patients treated for skin damage:

  * Diffuse skin sclerosis (rising above the elbows and / or knees)
  * First clinical sign of systemic sclerosis outside of Raynaud's phenomenon going back less than three years
  * Failure to take other concomitant immunosuppressive treatments or in the last 3 months except corticosteroids.
* In patients treated for lung damage:

  * Interstitial lung damage identified on chest CT, chest x-ray
  * Any duration of progression of systemic scleroderma
  * Prescription of MMF in first line or in relay of a treatment with Cyclophosphamide.
  * Absence of biotherapy in the last 6 months.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving MMF for another indication than skin or lung damage to systemic sclerosis (after lung transplantation for example).
  * Contraindication to MMF: Hypersensitivity to the product. Pregnancy.
  * In patients treated for skin damage:
    * Failure to take other concomitant immunosuppressive treatments or in the last 3 months except corticosteroid therapy.
    * No treatment with biotherapy in the last 6 months
  * In patients treated for lung damage:
    * No treatment with biotherapy in the last 6 months
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Skin efficacy | 1 year
  Modified Rodnan skin score (mRSS) : min 0 max 51. A diminution in the mRSS of more than 25% from the initial value was considered as improved. On the contrary, an increase in the mRSS over 25% was considered as deteriorated. All other variations of mRSS were classified as stable. Minimal clinically important difference was also tested (worsening of mRSS ≥ 4.7).

SECONDARY OUTCOMES:
Pulmonary efficacy.1 | 1 year
  Modification in FVC
Pulmonary efficacy.2 | 6 months and 1 year
  Modification in DLCO

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin hospital, AP-HP, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Gelder T, Le Meur Y, Shaw LM, Oellerich M, DeNofrio D, Holt C, Holt DW, Kaplan B, Kuypers D, Meiser B, Toenshoff B, Mamelok RD. Therapeutic drug monitoring of mycophenolate mofetil in transplantation. Ther Drug Monit. 2006 Apr;28(2):145-54. doi: 10.1097/01.ftd.0000199358.80013.bd. PMID 16628123
- [Background] Zahr N, Arnaud L, Marquet P, Haroche J, Costedoat-Chalumeau N, Hulot JS, Funck-Brentano C, Piette JC, Amoura Z. Mycophenolic acid area under the curve correlates with disease activity in lupus patients treated with mycophenolate mofetil. Arthritis Rheum. 2010 Jul;62(7):2047-54. doi: 10.1002/art.27495. PMID 20506558
- [Background] Chaigne B, Gatault P, Darrouzain F, Barbet C, Degenne D, Francois M, Szymanski P, Rabot N, Golea G, Diot E, Maillot F, Lebranchu Y, Nivet H, Paintaud G, Halimi JM, Guillevin L, Buchler M. Mycophenolate mofetil in patients with anti-neutrophil cytoplasmic antibody-associated vasculitis: a prospective pharmacokinetics and clinical study. Clin Exp Immunol. 2014 May;176(2):172-9. doi: 10.1111/cei.12246. PMID 24304103